CLINICAL TRIAL: NCT00731861
Title: Phase I, Pharmacokinetic, Pharmacodynamic Trial of PTK787 and Paclitaxel in Combination for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0412-21/ IUCRO-0101
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Neoplasm Metastasis; Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma | interventions — Paclitaxel; vatalanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Paclitaxel plus PTK787
  Interventions: Drug: Paclitaxel plus PTK787

INTERVENTIONS:
Drug: Paclitaxel plus PTK787 — Paclitaxel will be given on days 1 and 15 over 28 days in cycle 1 with PTK787 on days 3 to 28. PTK787 WILL BE TAKEN AT NIGHT.
  In cycle 2 and beyond, paclitaxel will be given on days 1, 8 and 15 every 28 days . PTK787 will be taken orally NIGHTLY.

SUMMARY:
This study will evaluate PTK787, a new oral drug that stops blood vessel development, in combination with Paclitaxel in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically confirmed malignancy that is unresponsive to curative therapy and for which no conventional therapy exists
* ECOG Performance Status 0-2
* Measurable or evaluable disease
* Laboratory values within protocol limits within 2 weeks prior to registration
* Life expectancy ≥ 12 weeks
* Patient or guardian must have written informed consent obtained according to local guidelines
* Women of child-bearing potential (non-sterile) must use appropriate barrier contraception for duration of study (negative pregnancy test required at baseline). Oral contraceptives will not be an acceptable form of contraception
* Patients may have received prior standard taxane therapy, but have never progressed on taxane-based therapy.

Exclusion Criteria:

* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis).
* Prior chemotherapy ≤ 3 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
* Prior biologic or immunotherapy ≤ 2 weeks prior to registration. Patients must have recovered from all therapy-related toxicities
* Prior full pelvic field radiotherapy ≤ 4 weeks or limited field radiotherapy ≤ 2 weeks prior to randomization.
* Major surgery (i.e., laparotomy) ≤ 4 weeks prior to randomization. Minor surgery ≤ 2 weeks prior to randomization.
* Patients who have received investigational drugs ≤ 4 weeks prior to registration
* Prior therapy with anti-VEGF agents
* Peripheral neuropathy with functional impairment ≥ CTC grade 2 neuropathy, regardless of causality
* Pleural effusion or ascites that causes respiratory compromise (≥ CTC grade 2 dyspnea)
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not employing an effective method of birth control.
* Patient agrees to avoid grapefruit (juice and fruit)

Any of the following concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study:

* Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
* Unstable angina pectoris
* Congestive heart failure greater than NYHA classification ≥ Grade 1 (can be controlled with medication)
* Myocardial infarction ≤ 6 months prior to registration and/or randomization
* Serious uncontrolled cardiac arrhythmia
* Uncontrolled diabetes at discretion of investigator
* Active or uncontrolled infection requiring intravenous antibiotics
* Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* Patients at risk of QT prolongation such as patients with congenital long QT syndrome or with long QTc at baseline (i.e. QTc greater than 450 msec in males, and greater than 470 msec in females) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-05; Primary Completion 2008-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of escalating doses of paclitaxel in combination with PTK787 | Baseline through End of Study

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of paclitaxel alone and in combination with PTK787 from patients with cancer accrued to this study | Baseline through End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Chiorean, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States